CLINICAL TRIAL: NCT00161200
Title: Studies of Esophageal Metaplasia Using a Novel Antibody: Reversibility of Columnar Metaplasia by Proton Pump Inhibitor
Brief Title: Esophageal Metaplasia Using a Novel Antibody: Reversibility by Proton Pump Inhibitor
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4310; 120303 (Other: CINJ); NIH 1R01 DK3618-01
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Esophageal Metaplasia
Keywords: Esophageal Metaplasia
MeSH Terms: interventions — Ranitidine; Pantoprazole

INTERVENTIONS:
Drug: Ranitidine & Pantoprazole

SUMMARY:
In this project, we are trying to identify patients with the earliest signs of abnormality in the lining of the lower part of the food pipe (or esophagus) known as intestinal metaplasia (IM); also commonly called Barrett's esophagus or Barrett's Epithelium (BE). IM is sometimes difficult to diagnose by routine microscopic examination (called histology). We have developed a specific antibody, a protein called immunoglobulin that specifically reacts with another partner protein, if it exists. Using this marker antibody (called mAb Das-1) that has been patented (US patent #5,888,743), we have shown that this marker can detect the abnormal changes in the distal esophagus before it is evident by histology. IM usually develops in the face of long-term acid reflux from the stomach to the esophagus and causes the lining to change from the normal squamous type (like that of skin) to a type of lining normally seen in the small intestine and colon. A subgroup of patients with IM may, subsequently, develop histologically evident Barrett's Epithelium and a small percent of these patients may develop cancer of the esophagus. Thus, BE is considered as a pre-cancerous condition. We already have an ongoing IRB for the portion of the project involving taking biopsies and performing the antibody staining to identify patients that react with the antibody but histologically negative for BE.

DETAILED DESCRIPTION:
We propose to study prospectively 68 patients who have been identified as positive with mAb DAS-1 immunostaining without histological evidence of specialized columnar epithelium ("True Barrett's" epithelium) during routine endoscopy for dyspepsia or GERD symptoms. These patients have been studied for initial screening for antibody staining under IRB protocol #1698. This number is based on the statistical analysis by Fisher's exact test and has 90% power to detect a 30% negativity (mAb Das-1 positive to negative) at a p<0.05 level. During participation in IRB Protocol #1698, initial biopsy specimens were taken at:

* the squamo-columnar junction (at least 2 sites - 12 o'clock and 6 o'clock positions and any other area with mucosal "tongues" of columnar epithelium),
* one from squamous epithelium at the distal esophagus to seek for the presence of esophagitis,
* one from antrum for the presence or absence of intestinal metaplasia of the stomach,
* and one from the gastric cardia.

Following endoscopy and participation in IRB Protocol #1698, for the symptomatic patients who are not taking any proton pump inhibitor, an H2 blocker, Ranitidine (ZantacÒ) 150 mg twice daily, will be started while the biopsy is being analyzed for histology and immunocytochemical stainings. This is usually completed within 2 weeks. Patients who showed positive reactivity in at least one biopsy sample taken during participation in Protocol #1698 with mAb Das-1 will be included in this study. Patients who have been taking a proton pump inhibitor (PPI) for longer than 3 months preceeding study entry are not eligible to participate in this study. Patients who have been taking proton pump inhibitors for 3 months or less at the time of the endoscopy and biopsy screening for mAb Das-1, may participate in this study 4 weeks after discontinuing the PPI (i.e., a 4 week washout period).

Patients will be randomized in a double-blinded fashion to receive either Pantoprazole, 40 mg twice daily (34 patients), or continued on Ranitidine, 150 mg twice daily (34 patients) for a total period of 6 months. Pantoprazole and Ranitidine will be provided by Wyeth and the code will be kept by the pharmacy department at The Cancer Institute of New Jersey. The drugs will be provided free of cost to the patients for the entire period. Patients will be followed as out-patients at three-month intervals up to 6 months. Patients will be advised to return any unused capsules during the follow-up visits. The number of unused capsules as well as review of the patient's medication diary will allow assessment of non-compliance. Patients must be at least 75% compliant to remain on the study. If any patient complains of persistent symptoms, an effort will be made to provide relief with antacids, as much as needed. However, if the patient is still symptomatic, they will be taken off the study and unblinded. If the patient is on Ranitidine they will be switched to open label Pantoprazole and will be followed and further treated in a routine manner. If the patient is taking Pantoprazole, pH monitoring to document acid reflux and planning of further management will be determined.

All patients will have a follow-up endoscopy at 6 months, with no cost to the patient. This cost will be born by the grant received by Dr. Das. Additional endoscopy will be performed at 12 months and 24 months, which is the current "standard care" procedure for surveillance in such patients. Follow-up biopsy specimens will be taken the same way as the initial specimens and processed to see any changes in histology and mAb Das-1 reactivity.

ELIGIBILITY:
Inclusion Criteria:

* Dyspeptic symptoms, upper abdominal pain, heartburn, regurgitation;
* Endoscopically - normal appearing GE junction, irregular z-line, or erosive esophagitis up to Grade 2.

Exclusion Criteria:

* Barrett's esophagus (Endoscopically greater than 2 cm of columnar epithelium on endoscopy and the presence of specialized columnar epithelium on histology);
* Patients who have been taking a PPI longer than the 3 months proceeding study entry. Patients currently taking a PPI but for less than 3 months who are not willing to discontinue PPI treatment for 4 weeks prior to enrollment into this study.
* Severe esophagitis Grade 3 or 4
* Documented active duodenal or gastric ulcer (at least 0.5cm diameter). Patients with erosions can be included.
* Presence of esophageal varices
* History of gastric surgery altering normal anatomy (eg, Billroth procedure, gastric bypass)
* Pregnant or nursing patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-12; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
The monoclonal antibody mAb Das-1 has been shown to react with a colonic epitope that is expressed in Barrett's Esophagus. Recent work has shown that it may be able to detect the changes of Barrett's Esophagus before it is histologically evident. In

CONTACTS AND LOCATIONS:
Overall Officials: Kiron Das, MD, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Cancer Institute of New Jersey, New Brunswick, New Jersey, United States